CLINICAL TRIAL: NCT04623268
Title: Detecting Abdominal Aortic Aneurysms in First Degree Relatives (Adult Offsprings) to AAA Patients (DAAAD)
Acronym: DAAAD
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Rebecka Hultgren, Professor, adjunct, Karolinska University Hospital
Other Study IDs: DAAAD
Record Dates: First submitted 2020-10-02; First posted 2020-11-10 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult offspring: Adult female and male offspring to AAA patients 45-80 years of age at inclusion Children to detected AAA patients. Found in the Multigeneration registry
  Interventions: Diagnostic Test: Ultrasound and questionnaire
- Control group: Matched women and men, without parents with AAA. Matched in the Swedish Multigeneration registry
  Interventions: Diagnostic Test: Ultrasound and questionnaire

INTERVENTIONS:
Diagnostic Test: Ultrasound and questionnaire — One invititation to identified adult offspring to have an ultrasound to detect an AAA. The prevalence in this Group (strata for sex) will be compared to a random selected matched Control group

SUMMARY:
The 8-12 fold higher risk for sisters and brothers of patients with Abdominal Aortic Aneurysms (AAA) to develop AAA compared to persons in the population is well known in the scientific community. Recently the value of the screening program for siblings has been analyzed and is shown to be highly cost-efficient, similar to the population based screening of 65-year old men for AAA. Most importantly detection of siblings also adresses and includes women at risk. The adult offsprings to AAA patient would hypothetically bear the same risk of AAA as siblings. This has never been evaluated scientifically due to the practical difficulties in tracking the offspring and inviting them to screening at an age when they are at risk of AAA-disease. In Sweden, the unique multigeneration registry exists which could support such detection, with the possibility to track adult offspring to patients, and investigate the true contemporary prevalence in them.

The DAAAD project aims at investigating the prevalence in adult offspring parallel to developing a model for such a selective screening program

DETAILED DESCRIPTION:
This project will evaluate four questions

1. Feasibility of study design; can we evaluate the prevalence of AAA by inviting and detecting risk groups in national registries ?
2. Point prevalence of AAA in a riskgroup of adult offspring to AAA patients as compared to a matched control group
3. Quality of Life in risk groups: measuring HADS, EQ-5D and questionnaire on heredity, including their awareness on their risk for AAA
4. Cost-effectiveness of such a national program based on prevalence and EQ-5D

This program will evaluate the risk for AAA in adult offspring and also evaluate a highly probable effective registry-based detection route. This could be more cost-efficient than any other AAA screening program, since the prevalence presumably is very high, and the registry-based route could be cheaper than nurse-based detection or incidental screening. The ultimate benefit of this program will be a crude reduction of sudden deaths from AAA for adult offspring to AAA patients, and this will be specifically impressive for the female relatives that are never subjected to any AAA-screening in our country.

ELIGIBILITY:
Inclusion Criteria:

Adult offspring to registered AAA parent (adult offspring) adult offspring not having a AAA parent (Controls)

-

Exclusion Criteria:

Not living in Stockholm below 45 or above 80

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Stratified analysis
Study Population: Random selection of Adult offspring to registered AAA parent (adult offspring) and adult offspring not having a AAA parent (Controls)
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of AAA | baseline
  Ultrasound or CT 30 mm aortic diameter

SECONDARY OUTCOMES:
Awareness of hereditability and anxiety levels | baseline
  Questionnaire based information

OTHER OUTCOMES:
Feasibility of registry-based detection model for screening. | One year after baseline
  Comparison can be made with the screening program in men. The outcome here is to explore if it is possible to implement this register model nationally at reasonable cost and work load. Participation rates, detailed analysis of non-participants in the risk group vs control group. Screening models are measured as feasible if participation >50%.
Cost Effectiveness of program measured by quality-adjusted life-years | One year after baseline
  Quality-adjusted life-years (QALYs) The prevalence in adult offspring, including cost of program, gives cost-effectiveness, probability of cost-effectiveness at different willingness-to-pay (WTP) thresholds, reduction in AAA death gained and total costs on a national scale. Presented as QUALY.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecka Rebecka, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Cannot share with patients' ID due to Ethic board regulation

REFERENCES:
- [Derived] Fattahi N, Linne A, Roy J, Stenman M, Svensjo S, Nilsson O, Hultgren R. Prevalence of abdominal aortic aneurysm (AAA) in first-degree relatives: detecting AAA in adult offspring of AAA patients. BJS Open. 2024 Jan 3;8(1):zrad163. doi: 10.1093/bjsopen/zrad163. PMID 38195162
- [Derived] Hultgren R, Fattahi N, Nilsson O, Svensjo S, Roy J, Linne A. Evaluating feasibility of using national registries for identification, invitation, and ultrasound examination of persons with hereditary risk for aneurysm disease-detecting abdominal aortic aneurysms in first degree relatives (adult offspring) to AAA patients (DAAAD). Pilot Feasibility Stud. 2022 Dec 12;8(1):252. doi: 10.1186/s40814-022-01196-9. PMID 36503690

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04623268/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04623268/ICF_000.pdf